CLINICAL TRIAL: NCT00359216
Title: A Double-Blind Placebo-Controlled, Randomized, Parallel-Group, Single-Site Study of Mometasone Furoate Nasal Spray (MFNS) In Subjects With Sleep-disordered Breathing Associated With Perennial Allergic Rhinitis (PAR) Using Home-Monitored Cardio-Respiratory Methodology.
Brief Title: The Effects of Mometasone Furoate Nasal Spray in Subjects With Sleep-disordered Breathing (SDB) Associated With Perennial Allergic Rhinitis (Study P04726)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04726
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Perennial Allergic Rhinitis; Obstructive Sleep Apnea; Sleep Disorder
Keywords: Hypopnea Syndrome
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Sleep Apnea, Obstructive; Sleep Wake Disorders | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mometasone furoate nasal spray (Experimental)
  Interventions: Drug: Mometasone furoate nasal spray
- Placebo nasal spray (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate nasal spray — MFNS, 50 mcg/spray. Each subject to take 200 mcg (4 sprays) once daily in the morning.
  Other Names: Nasonex
  Arms: Mometasone furoate nasal spray
Drug: Placebo — Placebo nasal spray. Each subject to take 4 sprays once daily in the morning.
  Arms: Placebo nasal spray

SUMMARY:
This is a Phase 4 randomized, placebo-controlled, parallel-group, single-center, double-blind study to evaluate the effects of mometasone furoate nasal spray (MFNS) in subjects with Sleep-disordered Breathing (SDB) associated with perennial allergic rhinitis (PAR) using Peak Nasal Inspiratory Flow (PNIF), Embletta device home-monitored cardiopulmonary evaluations, and rhinitis evaluations and questionnaires. Approximately 30 subjects 18 to 60 years of age with symptomatic PAR (with or without SAR) will be selected and randomized at one study site. The anticipated duration of subject participation in the study is approximately 39 days. Subjects who qualify at the Screening Visit will complete a 10-14 day run-in/screening period. Following the run-in period, subjects who meet the qualifications at the Baseline Visit will be treated with study medication for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Demonstration of willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Ages 18 to 60 years, of either sex, and of any race.
* A 2-year or longer history of perennial allergic rhinitis (PAR) with or without SAR.
* Skin test positive to a relevant prevalent perennial allergen or seasonal allergens if the subject also has SAR done either at the Screening Visit or within the previous 12 months.
* At the Screening Visit (Visit 1) subject must have TNSS of >=12 our of a possible 24, nasal congestion score of 4 out of a possible 6 on congestion, an Interference With Sleep average score of (2) moderate over 7 nights prior to the Screening Visit.
* At the Baseline Visit (Visit 2) scores, reflective over the previous 12 hours, of 4 or more for nasal congestion using a categorical whole-number symptom severity scale encompassing 7 severity ratings on at least 6 of the 15 recordings of the Run-in period which may include the morning of the Baseline Visit (Visit 2).
* At the Baseline Visit (Visit 2) subject must have a TNSS of more than >=12 out of a possible 24 reflective over the past 12 hours on at least 6 or more of the 15 recordings of the Run-in period, which may include the morning of the Baseline Visit.
* Current complaint of sleep disturbance while symptomatic with PAR and have a score of at least 2 with the Interference with Sleep scale on at least 4 out of the 8 AM diary recordings during the Run-in period and may include the morning of Visit 2 (Baseline).
* The number of AH events per hour will be recorded but should not exceed 30 per hour.
* Freedom from any clinically significant disease (other than PAR or SAR) that would interfere with the study evaluations.
* Confirmation by subject that he/she is practicing adequate contraception: Female volunteers of childbearing potential (including women who are less than 1 year postmenopausal and women who will be sexually active during the study) must agree to use a medically accepted method of contraception or be surgically sterilized prior to screening and while receiving protocol-specified medication. Women who are postmenopausal for >1 year (ie, women who have experienced 12 consecutive months of amenorrhea) will be exempted from the use of contraception during the study. Acceptable methods of contraception include condoms (male and female) with or without a spermicidal agent, diaphragm or cervical cap with a spermicidal agent, medically prescribed intrauterine device (IUD), oral or injectable hormonal contraceptives, and surgical sterilization (eg, hysterectomy or tubal ligation).
* Understanding of, and ability to adhere to, the dosing and visit schedules, and agreement to record symptom severity scores, medication times, concomitant medications, and adverse events accurately and consistently in a daily diary.

Exclusion Criteria:

* Pregnant or intention to become pregnant during the study
* Breast-feeding or intention to breast-feed during the study or within 30 days after study completion
* Currently medication for PAR, or during the 10 days prior to the Screening Visit, treatment for SAR or PAR with an antihistamine or a nasal inhaled corticosteroid.
* Current or a history of frequent (2 or more episodes per year for the past 2 years) clinically significant sinusitis or chronic purulent postnasal drip.
* Recent nasal septum ulcers, nasal surgery, or nasal trauma; postpone inclusion until healing has occurred.
* A diagnosis of rhinitis medicamentosa.
* Upper or lower respiratory tract or sinus infection that required antibiotic therapy with the last dose 14 days prior to screening, or a viral upper or lower respiratory infection within 7 days prior to screening.
* Nasal structural abnormalities, including large nasal polyps and marked septum deviation, that significantly interfere with nasal airflow.
* Bronchial asthma that cannot be controlled by short-acting beta 2-agonist adrenergic receptor agonists.
* Current desensitization immunotherapy and expectation of receiving an increase in dose during the study. Subject may not receive desensitization treatment within 24 hours prior to a study visit.
* Failure to observe the designated washout periods for any of the prohibited medications outlined in section 6.2 of the protocol.
* Previous randomization into the study.
* Current evidence of clinically significant hematopoietic, cardiovascular, hepatic, immunologic, renal, neurologic, psychiatric, autoimmune disease, or other disease that precludes the subject's participation in the study, or the subject's ability to complete the diary cards.
* Active or quiescent tuberculosis infection of the respiratory tract, untreated fungal, bacterial, or systemic viral infections, or ocular herpes simplex.
* Compromised ability to provide informed consent.
* A history of non-compliance with medications or treatment protocols.
* Morbidly obese (BMI >= 40).
* Night-shift working schedule with no standard asleep at night/awake during the day cycle.
* Any clinically significant deviation from the appropriate reference range in the physical examination that, in the investigator's judgment, may interfere with the study evaluation or affect subject safety.
* a situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Participation in any other clinical study(ies).
* Subject is on the staff, affiliated with, or a family member of the staff personnel directly involved with this study.
* Subject is allergic to or has sensitivity to the study drug or its excipients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meltzer EO, Munafo DA, Chung W, Gopalan G, Varghese ST. Intranasal mometasone furoate therapy for allergic rhinitis symptoms and rhinitis-disturbed sleep. Ann Allergy Asthma Immunol. 2010 Jul;105(1):65-74. doi: 10.1016/j.anai.2010.04.020. PMID 20642206

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a screening period followed by a 7-day run-in period, followed by the treatment period.
Groups:
- Mometasone Furoate Nasal Spray: 100 mg of suspension provided 50 mg of mometasone furoate monohydrate. Subjects were instructed to administer 2 sprays into each nostril every morning. The total dosage of 4 sprays (2 per nostril) thus provided 200 mg daily to subjects receiving active drug. Treatment was to be administered for a nominal period of 28 days, to a maximum of 32 days.
- Placebo Nasal Spray: The placebo nasal spray was identical in appearance to the active MFNS. The composition was identical to the commercial formulation, an aqueous suspension without the active ingredient (mometasone furoate monohydrate). The administration was identical to MFNS.
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Started | 20 | 10
Completed | 20 | 9 (Completed treatment but simultaneously partaking in other study,final study procedures not performed)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 10 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.55 (10.11) | 33.70 (8.11) | 34.27 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index
Description: Apnea-Hypopnea Index (AHI), used to assess severity of sleep apnea based on total number of complete cessations (apnea) and partial obstructions (hypopnea) of breathing occurring per hour of sleep. Determined by the frequency of occurrence of apnea-hypopnea episodes measured during sleep at home by an Embletta device.
Time Frame: change from baseline (screening) at the end of 28 days of treatment
Population: Diary data over interval of days was derived using the mean of non-missing entries. No imputation was applied to any other missing data
Measure: Mean (Standard Deviation); unit: apnea-hypopnea episodes per hour
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 20 | 9
apnea-hypopnea episodes per hour | 1.0 (2.1) | 1.6 (3.8)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; The p-value is obtained by F-test in ANCOVA to assess the treatment group difference in changes from baseline, adjusted for baseline; Test type: Superiority or Other; p = 0.9219, ANCOVA

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate Nasal Spray | Placebo Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (N=20) | Placebo Nasal Spray (N=10)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less